CLINICAL TRIAL: NCT04797481
Title: Pilot Testing of an Online Rehabilitation Intervention Aiming to Support People With Heart Failure.
Brief Title: Pilot Testing of an Online Rehabilitation Intervention for People With Heart Failure (PORIAS-HF).
Acronym: PORIAS-HF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: King's College London (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ER30631161
Record Dates: First submitted 2021-03-04; First posted 2021-03-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel Intervention (Experimental): Novel Intervention Exercise group.
  Interventions: Procedure: Exercise
- Control (Active Comparator): Self-managed Exercise group.
  Interventions: Procedure: Self-managed exercise

INTERVENTIONS:
Procedure: Exercise — Group A participants will be invited to attend up to 24 exercise sessions (2 sessions per week and a 3rd optional) and 2 virtual (online; a 3rd will be optional) HF workshops over 8 weeks. All sessions will be delivered via online platforms, with 1 facilitator supporting up to 8 participants simultaneously in each session.
  Arms: Novel Intervention
Procedure: Self-managed exercise — Group B participants will be provided with a self-care exercise programme. The exercise programme will be home-based with a mixture of online video calls and telephone support contacts, alternating once every other week. The video or telephone contacts will be mutually agreed by the patient and the facilitator at a mutually convenient time and will aim to support Group B participants, by offering advice and tracking progress. Patients will be provided with two exercise programmes: I) a chair-based exercise programme (DVD will be provided), and ii) a progressive walking training programme (a manual will be provided). Patients will be advised to exercise ≥3 times per week, starting from their own personal level and gradually building up over 8 weeks in session's duration, frequency of sessions per week, and walking pace.
  Arms: Control

SUMMARY:
The inability of the heart to pump out blood to the rest of the body organs is called heart failure (HF). HF affects almost 920,000 people in the UK, costing the NHS up to £2.33bn/year. Physical exercise programmes aiming to improve the heart's ability to pump out blood are used to a) reduce the risk of life-threatening events (e.g., heart attack), b) reduce admissions to hospital and c) improve individual's physical independence (e.g., walking unsupported, being able toperform daily essential activities). However, these physical exercise programmes have been cut short under the current COVID-19 pandemic, with support in most UK regions being restricted to online videos and advice. With many people with HF being asked to be "shielded" or "self-isolate" for an unknown duration, it is important to develop a reliable and cost-effective physical exercise service to support this clinical group. The research team has developed a novel physical exercise programme, fully-delivered online. Before assessing if it could improve clinical outcomes (e.g., heart's ability to pump out blood) and how cost-effective it could be, a 10-month pilot study is proposed that will assess if the proposed online physical exercise programme could be performed in people with HF. Thirty participants will be allocated at random into two groups: Group A will receive up to 24 exercise sessions and up-to 3 lifestyle workshops, in addition to usual care over a 2-month period. Group B will receive a self-care exercise programme (≥3 sessions per week) for a two-month period in addition to usual care. Prior to the group random allocation, online assessments will be performed including demographics and clinical history, the ability to perform daily activities, sedentary or physical activity habits and quality of life. The assessments including interviews to assess participant's experiences will be repeated at 2 months

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs. of either gender
* Confirmed diagnosis (by echocardiography) of HF reduced left ventricular ejection fraction
* Sinus rhythm N-Terminal pro-Brain Natriuretic Peptide (NTproBNP) is >400 ng/L at the time of referral to the diagnostic clinic if in sinus rhythm.
* Ability to exercise

Exclusion Criteria:

* Non-ambulant status
* Current pregnancy
* Scheduled major cardiac surgery
* The presence of an ICD or CRT-D device
* Severe pulmonary hypertension defined as systolic PAP of >60 mmHg
* NYHA function class IV
* Lack of internet connection
* Inability/unwillingness to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Adherence | 2 months
  Number of sessions completed.
Acceptability of procedures. | 2 months
  Acceptability of procedures will be assessed by examining reasons for drop-out in discontinuing participants and comparing attrition between groups
Recruitment rates. | 2 months.
  Recruitment rates will be measured as rate of invited participants who are eligible and consenting

SECONDARY OUTCOMES:
30-second chair-stand test | Baseline.
  30-second chair-stand test
30-second chair-stand test | 2 months
  30-second chair-stand test
Step in place test | Baseline
  Step in place test (2mins)
Step in place test | 2 months
  Step in place test (2mins)
arm curl test | baseline
  arm curl test
arm curl test | 2 months
  arm curl test
EQ5D-5L | baseline
  The EQ5D-5L questionnaire will be completed, to support assessment of quality of life.
EQ5D-5L | 2 months
  The EQ5D-5L questionnaire will be completed, to support assessment of quality of life.
MLHFQ | Baseline.
  The MLHFQ questionnaire will be completed, to support assessment of quality of life.
MLHFQ | 2 months
  The MLHFQ questionnaire will be completed, to support assessment of quality of life.
BREQ-2 | Baseline.
  The BREQ-2 questionnaire will be completed, to support assessment of quality of life.
BREQ-2 | 2 months
  The BREQ-2 questionnaire will be completed, to support assessment of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Markos Klonizakis, D.Phil, Principal Investigator — Sheffield Hallam University
Locations (1):
- Sheffield Hallam University, Sheffield, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No